CLINICAL TRIAL: NCT01719198
Title: Usefulness of Fecal Calprotectin for Screening Colon Adenoma in Korean Population
Brief Title: Usefulness of Calprotectin for Colon Adenoma Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Chul Min Park, MD, clinical instructor, Konkuk University Medical Center
Other Study IDs: KUH1220
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Colon Adenoma
Keywords: adenoma; calprotectin
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool specimen
Oversight: Data Monitoring Committee: No

SUMMARY:
The fecal calprotectin assay is used widely for inflammatory bowel disease diagnosis and the assessment of the disease activity. Some adenoma patients have elevated fecal calprotectin level, which could mean the role of fecal calprotectin as a screening marker for colon adenoma. We will investigate the usefulness of fecal calprotectin as colon adenoma marker for screening in this study.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old adult population

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who visit KUH healthcare center for colonoscopy in Korea over 18 years old adult population
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
fecal calprotectin level | 1 day (at the hospital visit)

CONTACTS AND LOCATIONS:
Overall Officials: Yeo-Min Yun, MD, PhD, Principal Investigator — Konkuk University
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea